CLINICAL TRIAL: NCT01278108
Title: Double-blind, Placebo-controlled, Dose-ranging Trial for the Assessment of Safety, Tolerability, Pharmacokinetics (PK), and Pharmacodynamics (PD) of Single Ascending Oral Doses, and Multiple Oral Doses of GLPG0778 in Healthy Subjects.
Brief Title: First-in-Human Single Ascending and Multiple Dose of GLPG0778
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: GLPG0778-CL-101; 2010-023199-16 (EudraCT Number)
Record Dates: First submitted 2011-01-14; First posted 2011-01-17 (Estimated); Last update posted 2011-10-18 (Estimated); Status verified 2011-10

CONDITIONS: Healthy
Keywords: Safety; Tolerability; Pharmacokinetics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): single ascending doses
  Interventions: Drug: GLPG0778
- 2 (Placebo Comparator): single dose placebo
  Interventions: Drug: placebo
- 3 (Experimental): multiple dose, 7 days, capsules (dosing depends on outcome of single-dose part; can be once or twice daily).
  Interventions: Drug: GLPG0778
- 4 (Placebo Comparator): multiple dose, capsules, 7 days; scheme to match that of Study Arm 3.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: GLPG0778 — single ascending doses, oral solution (10 to 800 mg/dose) and capsules (100 mg/dose)
  Arms: 1
Drug: placebo — single dose, oral solution or capsule (matching corresponding study medication)
  Arms: 2
Drug: GLPG0778 — multiple dose, capsule, 7 days
  Arms: 3
Drug: placebo — multiple dose, capsule, 7 days
  Arms: 4

SUMMARY:
The purpose of the study is to evaluate the safety and tolerability of single ascending (SAD) and multiple (MD) oral doses of GLPG0778 compared to placebo (with and without food).

Also, pharmacokinetics (PK) and pharmacodynamics (PD) of GLPG0778 after single and multiple oral administration will be evaluated, and, if applicable, the maximum tolerated dose determined.

ELIGIBILITY:
Inclusion Criteria:

* healthy male
* body mass index (BMI) between 18-30 kg/m², inclusive.

Exclusion Criteria:

* any condition that might interfere with the procedures or tests in the study
* smoking
* drug or alcohol abuse

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-12; Primary Completion 2011-02 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of single and multiple dosing | up to 10 days postdose
  Tests will be performed to assess whether the study drug has any potentially adverse effect (laboratory tests on blood and urine for functioning of organs; cardiovascular testing, i.e. of heart and bloodcirculation). Also, participants will carefully be monitored by medical staff for vital signs, and asked to report any side effect experienced in the course of the study.

SECONDARY OUTCOMES:
Pharmacokinetics of single and repeated doses, including effect of food. | up to 10 days postdose
  Bloodsamples are taken on various timepoints to assess how much of the study drug is taken up in the blood (absorption), how long it stays in the blood (excretion), and whether any "breakdown"-products of the drug are present (metabolism).

CONTACTS AND LOCATIONS:
Overall Officials: Gerben van 't Klooster, PhD, Study Director — Galapagos NV; Lien Gheyle, MD, Principal Investigator — SGS Stuivenberg
Locations (1):
- SGS Stuivenberg, Antwerp, Belgium